CLINICAL TRIAL: NCT02470221
Title: Effect of Goal-Directed Intraoperative Fluid Therapy on Outcomes Following Laparotomy of Gynecological Malignancies and Orthopedic Surgery
Brief Title: Goal-directed Intraoperative Fluid Therapy in High-risk Surgery
Status: Completed | Type: Observational
Sponsor: Huang YuGuang (Other)
Responsible Party: Sponsor-Investigator, Huang YuGuang, Professor，Chairman, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: anesthesiologyPUMCH001
Record Dates: First submitted 2015-05-28; First posted 2015-06-12 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Complications; Fluid Overload
Keywords: goal-directed fluid therapy; intraoperative hemodynamics; postoperative complications
MeSH Terms: conditions — Postoperative Complications; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Goal-directed fluid therapy: The fluid in group Goal-directed fluid therapy will be administered based upon real-time monitoring stroke volume variation and cardiac output achieved by the Flo-Trac monitoring system.
  Interventions: Other: Applying goal-directed fluid therapy by continuous hemodynamic monitoring system
- Conventional fluid therapy: The fluid in group Conventional fluid therapy will be administered based on the principle crystalloid solution: colloid solution =2-3:1. The total volume of fluid will be adjusted in accordance with blood pressure, heart rate and urine output of each patient.
  Interventions: Other: Conventional fluid therapy

INTERVENTIONS:
Other: Applying goal-directed fluid therapy by continuous hemodynamic monitoring system — Applying continuous hemodynamic monitoring system ( Vigileo/Flotrac) to monitor Stroke Volume Variation and Cardiac Output and further manage intra-operative fluid therapy.
  Groups: Goal-directed fluid therapy
Other: Conventional fluid therapy — Applying conventional fluid therapy according to Peking Union Medical College Hospital standard.
  Groups: Conventional fluid therapy

SUMMARY:
This study is aim to assess the effect of goal-directed intraoperative fluid therapy on patient's postoperative incidence rates of complications, length of hospitalization and hospitalization cost.

This is an observational study followed cohort study design, due to the two therapies were not randomized assigned to the two cohorts. The details are described as follow.

DETAILED DESCRIPTION:
The study will be conducted in patients undergoing either elective laparotomy of gynecological malignancies or elective major orthopaedic surgery under prone position in Peking Union Medical College Hospital. The study included two stages.

In the first stage, one cohort of 300 participants with conventional fluid therapy will be involved, in which 150 patients will be selected with laparotomy of gynecological malignancies and150 patients will be selected with orthopedic surgery. All the participants in this stage will follow conventional fluid therapy to direct the amount of intraoperative fluid. Specifically, the fluid will be administered based on the principle crystalloid solution (colloid solution =2-3:1). The total volume of fluid will be adjusted in accordance with blood pressure, heart rate and urine output of each patient. It is a standard procedure in Peking Union Medical College Hospital. Then, the incidence of postoperative complications of each group will be recorded. In addition, sample size will be estimated based on above study's results (estimated 100 participants).

In the second stage, goal-directed therapy will be applied to another cohort of 300 participants, in which 150 patients undergoing laparotomy of gynecological malignancies and 150 patients undergoing orthopedic surgery. Specifically, the fluid will be administered based upon real-time monitoring stroke volume variation and cardiac output achieved by the Flo-Trac monitoring system. The incidence of postoperative complications of each group will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving elective laparotomy of gynecological malignancies (LGM): including cytoreductive surgery of ovarian cancer, radical hysterectomy and staging surgery of endometrial cancer ;
2. Major elective orthopedic surgery (OS): including spinal surgery, revision surgery of hip joints ;
3. Age ≥18 years, American Society of Anesthesiologists physical status I ～IV;
4. No arrhythmia;
5. Receiving general anesthesia;
6. Requiring monitoring of direct blood pressure due to the comorbidities of patients and the nature of surgical procedures.

Exclusion Criteria:

1. Emergent surgery;
2. Patients with aortic regurgitation;
3. Patients with aortic stenosis, peripheral arterial diseases or other diseases contradicting to arterial canalizations;
4. Patients with mental disorders or low intelligence quotient; patients who cannot cooperate or refuse to sign the consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent either laparotomy of gynecological malignancies or orthopedic surgery
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-02-10 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 30 days after the surgery
  the incidence of complications related to surgeries 30 days postoperatively. The complications include pneumonia, pulmonary embolism, cardiovascular events (myocardial infarction, heart failure), wound infection, gastrointestinal bleeding,nausea and vomitting，postoperative hemorrhage, ileus, deep venous thrombosis, cerebral infarction, cerebral embolism, cerebral hemorrhage, renal insufficiency and failure. Those complications are defined strictly to the reference published in 2009 New England Journal of Medicine （N Engl J Med. 2009 Oct 1;361:1368-75）

SECONDARY OUTCOMES:
hospital length of stay | participants will be followed for the duration of hospital stay, an expected average of 10 days
  the length of stay in hospital，from the hospitalized date to the leave date
hospital expenses | 30 days after the surgery
  total cost in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD, Study Chair — Peking Union Medical College Hospital

REFERENCES:
- [Background] Cecconi M, Fasano N, Langiano N, Divella M, Costa MG, Rhodes A, Della Rocca G. Goal-directed haemodynamic therapy during elective total hip arthroplasty under regional anaesthesia. Crit Care. 2011;15(3):R132. doi: 10.1186/cc10246. Epub 2011 May 30. PMID 21624138
- [Background] Kuper M, Gold SJ, Callow C, Quraishi T, King S, Mulreany A, Bianchi M, Conway DH. Intraoperative fluid management guided by oesophageal Doppler monitoring. BMJ. 2011 May 24;342:d3016. doi: 10.1136/bmj.d3016. PMID 21610051
- [Background] Wang P, Wang HW, Zhong TD. Effect of stroke volume variability- guided intraoperative fluid restriction on gastrointestinal functional recovery. Hepatogastroenterology. 2012 Nov-Dec;59(120):2457-60. doi: 10.5754/hge12283. PMID 22626878
- [Background] Ramsingh DS, Sanghvi C, Gamboa J, Cannesson M, Applegate RL 2nd. Outcome impact of goal directed fluid therapy during high risk abdominal surgery in low to moderate risk patients: a randomized controlled trial. J Clin Monit Comput. 2013 Jun;27(3):249-57. doi: 10.1007/s10877-012-9422-5. Epub 2012 Dec 22. PMID 23264068
- [Background] Donati A, Loggi S, Preiser JC, Orsetti G, Munch C, Gabbanelli V, Pelaia P, Pietropaoli P. Goal-directed intraoperative therapy reduces morbidity and length of hospital stay in high-risk surgical patients. Chest. 2007 Dec;132(6):1817-24. doi: 10.1378/chest.07-0621. Epub 2007 Oct 9. PMID 17925428
- [Derived] Che L, Zhang XH, Li X, Zhang YL, Xu L, Huang YG. Outcome impact of individualized fluid management during spine surgery: a before-after prospective comparison study. BMC Anesthesiol. 2020 Jul 22;20(1):181. doi: 10.1186/s12871-020-01092-w. PMID 32698766